CLINICAL TRIAL: NCT03966326
Title: Pectoralis and Serratus Nerve Blocks for Mastectomy: a Prospective, Randomized, Single-blind, Controlled Trial
Brief Title: Pectoralis and Serratus Nerve Blocks for Mastectomy: a Prospective, Randomized, Single-blind Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Preceptor of anesthesiology medical residency, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PECS II block
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain
Keywords: Mastectomy; (PECs) pectoral block
MeSH Terms: conditions — Pain, Postoperative | interventions — Sevoflurane; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Patients in placebo group will receive general balanced inhaled anesthesia with sevoflurane and fentanil
  Interventions: Drug: sevoflurane and fentanil
- PECS II group (Active Comparator): Patients in PECS II group will receive general balanced inhaled anesthesia with sevoflurane and fentanil
  Interventions: Drug: sevoflurane and fentanil plus PECS II block

INTERVENTIONS:
Drug: sevoflurane and fentanil — Patients will receive standard general anesthesia
  Other Names: Standard general anesthesia
  Arms: Placebo group
Drug: sevoflurane and fentanil plus PECS II block — Pacients will receive standard general anesthesia with sevoflurane and fentanil associated to PECS II block
  Other Names: Standard general anesthesia plus PECS II block
  Arms: PECS II group

SUMMARY:
Pectoral nerve block provides a good alternative to epidural or paravertebral block with a lower risk for the patient and that is shown as an optimal anesthetic option with reduction in postoperative pain, anesthetic and opioid consumption. The main objective of this study is to evaluate the quality of the perioperative analgesia of the PECS block in patients electively escalated for the accomplishment of mastectomy under general anesthesia.

DETAILED DESCRIPTION:
The advent of ultrasound made possible greater safety and the creation of new peripheral blocks that aim to reduce the morbidity of the anesthetic technique on the cancer patient. Pectoral nerve block (PEC Block) is technically simple and easily reproducible. Inspired by the infraclavicular approach, it aims at the anesthesia of the pectoral, intercostobrachial, intercostal III-IV-V-VI nerves and the long thoracic nerve 8 being a safe, reproducible technique with little discomfort for the patients, with few complications and allowing a good control of acute pain.

The hypothesis is that the realization of pectoral nerve block provides a good alternative to epidural or paravertebral block with a lower risk for the patient and that is shown as an optimal anesthetic option with reduction in postoperative pain, anesthetic and opioid consumption. Main objective is the evaluation of postoperative pain through opioid consumption in the first 24 hours postoperatively.

Patients will undergo a prospective, randomized, single blind, placebo controlled study in which the examiners responsible for the postoperative evaluation will not know which of the two groups were randomly assigned: 40 patients in the Control and 40 patients in the PECS Group . Patients will be randomized through a list generated by www.randomizer.org into two groups.

Patients will receive standard monitoring, pre-anesthetic medication with midazolam 0.05 mg / kg EV. All patients will receive balanced general anesthesia with fentanyl 2 mcg / kg, lidocaine 2 mg / kg, propofol 1-2 mg / kg, cisatracurium 0.15 mg / kg or Rocuronium 0.6 mg / kg. The PECS II group will receive an injection of 20mL of 0.5% Ropivacaine between the serratus and the smaller pectoralis and 10mL of 0.5% ropivacaine between the pectoralis major and minor muscles with the aid of ultrasonography. Maintenance of anesthesia in the two groups: general anesthesia balanced with sevoflurane (with and fraction expired from 1 to 3%, to maintain BIS between 40 and 60). Prophylaxis for postoperative nausea and vomiting will be performed with slow intravenous administration following the anesthetic induction of Dexamethasone 4 mg, and at the end of the surgery slow intravenous administration of Ondansetron 4 mg. At the end of surgery, patients in both groups will receive Dipyrone 2 g and Parecoxib 40 mg. Patients will be evaluated in the postoperative times: T1: arrival at the PACU, T2: 3 hours postoperatively or discharge from the PACU), T3: 12 hours postoperative, T4: 24 hours postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18 to 60 years, electively scheduled to perform mastectomy in the Base Hospital of the Federal District;
* Physical State 1, 2 or 3 the American Society of Anesthesiology (ASA);

Exclusion Criteria:

* Patients with unstable angina
* Patient with poorly controlled asthma
* Substance abuse
* Heart failure, greater than first degree atrioventricular block
* Pregnant women
* Patients with allergy to dipyrone, morphine;
* Patients with chronic pain;
* Patients with severe hepatic disease;
* Patients with severe kidney disease;
* Patients with neurological diseases;
* Included patients in other clinical studies currently or in the past three months under general anesthesia;
* Patients who refuse to participate in the study;
* Any other condition that, in the opinion of the investigator, may pose a risk to the patient or interfere with the study objectives;

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analogue Scale | Within the first 24 hours after surgery
  Quantify pain by Visual Analogue Scale (VAS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or un bearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonça, MD, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] O'Scanaill P, Keane S, Wall V, Flood G, Buggy DJ. Single-shot pectoral plane (PECs I and PECs II) blocks versus continuous local anaesthetic infusion analgesia or both after non-ambulatory breast-cancer surgery: a prospective, randomised, double-blind trial. Br J Anaesth. 2018 Apr;120(4):846-853. doi: 10.1016/j.bja.2017.11.112. Epub 2018 Feb 14. PMID 29576125
- [Derived] Mendonca FT, Nascimento LFC, Veloso NM, Basto GCP. Long-term Efficacy of Pectoserratus Plane Block (PSPB) for Prevention of Post-mastectomy Pain Syndrome: Extended Follow-up From a Randomized Controlled Trial. Clin J Pain. 2023 Jul 1;39(7):334-339. doi: 10.1097/AJP.0000000000001118. PMID 37083738